CLINICAL TRIAL: NCT03402295
Title: Superiority of the Triple Combinations of Bortezomib, Cyclophosphamide and Dexamethasone (VCD) Versus Cyclophosphamide, Thalidomide and Dexamethasone (CTD) in Patients With Newly Diagnose Multiple Myeloma, Eligible for Transplantation
Brief Title: Superiority of VCD Versus CTD in Patients With Newly Diagnose Multiple Myeloma Eligible for Transplantation
Acronym: GBRAM003r
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Responsible Party: Principal Investigator, Vania TM Hungria, Assintant Professor of Hematology oncology- Santa Casa de Sao Paulo Medical School, Grupo de Estudos Multicentricos em Onco-Hematologia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBRAM003r
Record Dates: First submitted 2017-12-28; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma; Effects of Chemotherapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Retrospectively compared two different groups of treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vcd- (Bortezomibe, cyclophosphamide and dexamethasone) (Active Comparator): Intervention - Bortezomib 1.3mg/m2 Intra venous or Subcutaneous once a week (D1-8-15-22) 35days cycle Intervention- Dexamethasone 40mg once a week for four weeks orally or Intravenously- total dose per cycle was 160mg.
  Intervention- Cyclophosphamide 900-2000mg- intravenously or orally- total dose monthly Total of four cycles
  Interventions: Drug: Bortezomib, cyclophosphamide, thalidomide, dexamethasone
- Ctd- Cyclophosphamide, thalidomide and dexamethasone (Active Comparator): Intervention- Cyclophosphamide 900-2000mg intravenously or orally total dose monthly Intervention- Thalidomide 100-200mg orally- daily dose Intervention -Dexamethasone 40mg once a week for four weeks each month- total dose per cycle was 160mg Total of four cycles (cycles of 28 each one)
  28 days each cycles- total of four cycles
  Interventions: Drug: Bortezomib, cyclophosphamide, thalidomide, dexamethasone

INTERVENTIONS:
Drug: Bortezomib, cyclophosphamide, thalidomide, dexamethasone — Comparison between two triple combination chemotherapy that include in different new drugs (bortezomibe e talidomida)
  Other Names: Velcade, genuxal, decadron

SUMMARY:
This study compared two main different induction protocols used to treat myeloma eligible patients in Brazil. VCD against CTD.

DETAILED DESCRIPTION:
The primary aim was observe response rate after 4 induction cycles.

ELIGIBILITY:
Inclusion Criteria:

* multiple myeloma newly diagnose elegible to autologous transplantation Patients submitted to ctd or vcd Myeloma patients newly diagnose >18yo

Exclusion Criteria:

* other chemotherapy induction protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2009-06-15; Primary Completion 2014-06-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Response rate better than very good partial response after 4 induction cycles | Response rate after induction phase - at the end of cycle 4- (28 days each cycle)- time frame trough study completion
  The primary outcome is to observe the difference response rate between VCD and CTD induction myeloma elegible patient

CONTACTS AND LOCATIONS:
Overall Officials: Edvan Cusoe, MD, Principal Investigator — Federal University of Bahia

IPD SHARING:
Plan to Share IPD: No